CLINICAL TRIAL: NCT04395378
Title: The Use of the Dexcom G6 in Commercial Pilots With Insulin Dependent Diabetes (DEXFLY)
Brief Title: Use of Dexcom G6 in Commercial Pilots With Insulin Treated Diabetes
Acronym: DEXFLY
Status: Suspended | Type: Observational
Why Stopped: COVID-19 policy of the University of Surrey
Sponsor: University of Surrey (Other)
Collaborators: UK Civil Aviation Authority (Unknown); Irish Civil Aviation Authority (Unknown); Austrian Civil Aviation Authority (Unknown)
Responsible Party: Sponsor
Other Study IDs: Spon_2019_015_FHMS
Record Dates: First submitted 2019-06-05; First posted 2020-05-20 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Flying pilots: Flying pilots holding class 1 and class 2 certificates
  Interventions: Device: Continuous Glucose monitoring DEXCOM G6

INTERVENTIONS:
Device: Continuous Glucose monitoring DEXCOM G6 — Continuous glucose monitoring during flight and normal living life

SUMMARY:
The investigators wish to explore the use of the CGMS Dexcom G6® in pilots with insulin-treated diabetes, who are flying commercial aircraft with Class 1 and flying instructors or private pilots with class 2 certificates.

The aim of this study is to explore the severity and number of hypoglycaemic episodes recorded with rtCGMS compared to the results from other self-glucose monitoring following the current protocol of the UK Civil Air Aviation (UKCAA), and to explore the possibility of the use of rtCGMS during flight and free living.

This will involve using CGM Dexcom G6® for continuous glucose monitoring for 6 months in flight time and during free living. The participants will be blinded for the results for the first month but will be encouraged to use the data from the CGMS Dexcom G6 ® for the following 5 months during the trial.

DETAILED DESCRIPTION:
People with diabetes sometimes consider that they are subjected to unfair discrimination in the occupational or work environment. These include safety-critical activities such as operating machinery and driving. Some occupations preclude the use of medications that lower blood glucose, particularly insulin. Safety regulators, occupational health physicians and national organisations frequently have to balance the competing priorities of individual rights against public safety.

Modern treatment, with advances in insulin therapy and glucose monitoring, combined with rigorous clinical assessment and review, has allowed stereotypical attitudes to be challenged, and advocated individual assessment with respect to safety criteria. Several national authorities (Australia, Canada, UK, and USA) have, over recent years, allowed private pilots to fly for recreation while receiving treatment with insulin Canada (in 2002) was the first country to allow commercial pilots, treated with insulin, to fly commercially and have granted licences to a small number of insulin-treated pilots on a case-by-case basis and subject to close supervision.

In 2010 the UK Civil Aviation Authority (CAA) convened an expert committee to review current scientific knowledge and international policies concerning flying. The committee advised that a protocol for safe flying could be developed and produced the first iteration with subsequent refinement. In 2012 the UK CAA started issuing Class 1 medical certificates for commercial flying to pilots with insulin-treated diabetes, having published a rigorous protocol and started collecting data systematically. Ireland and Austria have subsequently joined the protocol. The protocol has been shown to be feasible, practical and to date no safety concerns have arisen. The results from the first 26 pilots have been presented at the annual EASD conference and published in The Lancet Diabetes & Endocrinology .

ELIGIBILITY:
Inclusion Criteria:

* Any ethnithity
* Pilots requiring insulin replacement therapy
* Pilots holding a class 1 or class 2 certificate
* Pilots currently participating in the current scheme
* Able and willing to perform self-blood glucose monitoring.
* Able and willing to wear a Continuous Glucose Monitoring System (CGMS) for 6months

Exclusion Criteria:

* Outside of stated age range.
* Those who are part of the protocol but are not flying currently.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pilots with class 1 and flying instructors or private pilots with class 2 medical certificates with insulin dependent diabetes
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-12-05 (Actual); Primary Completion 2022-12-02 (Estimated); Study Completion 2022-12-02 (Estimated)

PRIMARY OUTCOMES:
Glucose concentration (mmol/L) | 18 months
  To compare the glucose monitoring CGMS Dexcom G6® with the usual self-glucose monitoring in pilots by way of assessing times achieved in safe Green flying range, in Amber flying range and in Red flying range as defined by the ARA.MED.330 diabetes protocol.

SECONDARY OUTCOMES:
Variability of glucose concentration (mmol/L) in-flight | 18 months
  Variability of glucose concentration while flying monitored using Dexcom G6 in comparison to the finger prick self-glucose monitoring
Variability of glucose concentration (mmol/L) at non-flying normal living | 18 months
  Time in and out of range during non-flying normal living (targets used as other clinical trials)
Quality of life (generic, disease-specific) evaluation and flying-specific evaluation scores. | 18 months
  Participants will be asked to fill in the quality of life (generic, disease-specific) evaluation and flying-specific evaluation questionnaires at the visit 1 and the end of the trial Visit 2.
HbA1c mmol/mol | 18 months
  HbA1C (mmol/mol) results from the participants' usual clinic visit at the CAA will be recorded in visit 1 and visit 2 .
Height (cm) | 18 months
  Height measured at the participants' usual clinic visit at the CAA will be recorded in visit 1 and visit 2
Weight (kg) | 18 months
  Weigh (kg) measured at the participants' usual clinic visit at the CAA will be recorded in visit 1 and visit 2
Blood pressure (systolic and diastolic) mmHg | 18 months
  Blood pressure (systolic and diastolic) mmHg measured at the participants' usual clinic visit at the CAA will be recorded in visit 1 and visit 2
Age (y) | 18 months
  Age of the participants' usual clinic visit at the CAA will be recorded in visit 1 and visit 2
Total Cholesterol (mmol/L) | 18 months
  Lipid profile values from the biochemical analysis obtained at the participants' usual clinic visit at the CAA will be recorded in visit 1 and visit 2
Creatinine (mmol/L) | 18 months
  Creatinine concentration from the biochemical analysis obtained at the participants' usual clinic visit at the CAA will be recorded in visit 1 and visit 2.
  This will be used to calculate glomerular filtration rate (GFR), mL/min/1.73 m2, or creatinine clearance using Cockcroft-Gault Equation.
Plasma albumin concentration (g/dL) | 18 months
  albumin concentration from the biochemical analysis obtained at the participants' usual clinic visit at the CAA will be recorded in visit 1 and visit 2. The ratio of will be used to calculate, the state of microalbumin urea in both visits.

OTHER OUTCOMES:
Glucose concentrations below 4 mmol/L | 18 months
  Incidence of hypoglycaemic episodes (all, minor, major and symptoms only) will be collected from Dexcom G6 monitoring and compare to the finger prick glucose values during the trial for 6 months.
Reactions to the sensors | 18 months
  Any adverse event such as discomfort to having the sensor under the skin and the adhesive covering the sensors during the trial will be recorded.
Aviation assessments as defined by the European Commission Aircrew Regulation ARA.MED.330 diabetes protocol. | 18 months
  Data collected from aviation assessments as defined by the European Commission Aircrew Regulation ARA.MED.330 diabetes protocol. This is a requirement for all pilots who fly on insulin.
Glucose concentration from the pilots log books for the previous 6 months | 18 months
  Glucose concentrations form the participating pilots' log books will be collected. the data will be analysed and compared to the data on the log books during the trial.

CONTACTS AND LOCATIONS:
Overall Officials: David Russell-Jones, BSc, Principal Investigator — University of Surrey
Locations (3):
- Diabetes Endocrinology General Internal Medicine,University of Graz, Graz, Austria
- Whitfield Clinic, Butlerstown North, Cork Rd, Waterford, Ireland
- Aviation house, Gatwick, West Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to identifiable data (e.g., name, address) will be limited to selected members of the research team and to regulatory authorities, the Sponsor, and the host organisation for auditing and monitoring purposes. This information and other personal details will not be included in analysis, or in publications or reports. All information collected during the study will be identified by a unique code so that the participant cannot be identified.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 18 months
Access Criteria: All data will be kept on secure CAA or University of Surrey computer servers and in a secure office environment within the CAA and University of Surrey.
  If data transfer is required password protected inscription will take place that meet the data transfer.

REFERENCES:
- [Derived] Garden GL, Shojaee-Moradie F, Hutchison EJ, Frier BM, Shaw KM, Heller SR, Koehler G, Mader JK, Maher D, Roberts GA, Russell-Jones DL. Continuous Glucose Monitoring by Insulin-Treated Pilots Flying Commercial Aircraft Within the ARA.MED.330 Diabetes Protocol: A Preliminary Feasibility Study. Diabetes Technol Ther. 2023 Aug;25(8):543-548. doi: 10.1089/dia.2023.0069. PMID 37384853